CLINICAL TRIAL: NCT05565612
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Effect of a Probiotic Mixture on Signs and Symptoms of Irritable Bowel Syndrome
Brief Title: Clinical Trial to Evaluate the Effect of a Probiotic Mixture on Signs and Symptoms of Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratorio Industrial de Herbodietetica Aplicada S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SII.PROB
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-10

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Pilot randomized, double-blind, placebo-controlled study of a duration of 12 weeks
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Normodigest Classic
  Multi-strain probiotic mixture (15 strains) with a concentration of 7,5 x 10^9 + fructooligosaccharides
  1 vial of 10 ml per day for 12 weeks
  Interventions: Dietary Supplement: Normodigest Classic
- Placebo group (Placebo Comparator): Maltodextrin-based placebo
  1 vial of 10 ml per day for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Normodigest Classic — Symbiotic composed of 15 probiotic strains and fructooligosaccharides as prebiotic
  Arms: Probiotic group
Dietary Supplement: Placebo — Compound based on maltodextrin and other excipients
  Arms: Placebo group

SUMMARY:
The clinical trial has a randomized, double-blind and placebo-controlled design, in which the effect of a probiotic mix wants to be evaluated, with a treatment of 12 weeks, in the evolution of the symptoms of Irritable Bowel Syndrome.

The 12 weeks of the treatment are structured in four in-person visits: Visit 1 (initial; week 0), Visit 2 (halfway; week 4), Visit 3 (halfway; week 8) and Visit 4 (final; week 12).

DETAILED DESCRIPTION:
Below, the four visits that compose the study and what to do in each one of them are described:

Visit 1 or initial (Week 0)

With the aim of recruiting patients, all patients diagnosed with irritable bowel who go to a consultation in the participant centres shall be informed of the study. If the patient shows interest, they shall be given detailed information about the study and the implications of their participation so that they can sign the informed consent if they wish so. Before signing, the patients shall have enough time to read and consider the detailed information and ask the investigator. The process of recruitment of patients shall continue until the sample size is reached.

Once the informed consent is signed, a doctor trained for the study shall make the initial interview in which the patient is tested to meet all the criterion for inclusion and none for exclusion (see clause 5.3.) and their clinical history.

The investigator shall proceed to assign to the patient the participant number on the study and, according to a previously elaborated randomization list, they shall be assigned the treatment that they shall receive during the study.

Once gotten to this point, the investigator shall value the severity and the symptoms of the Irritable Bowel Syndrome, by means of the IBS-SSS and IBS-QOL questionnaires (Annex I and II).

The patient shall be given the treatment with the assigned code, enough for the next programmed visit.

They shall be asked to turn in a stool sample and the nurse staff shall take a blood sample.

Visit 2 (Week 4) and visit 3 (Week 8)

In the halfway visits, in addition to value the symptoms of the disease with the scales detailed on the variable clause, the investigator shall register the adverse occurrences reported by the patient in a Case Report Form (CRF), as well as the concomitant treatments used.

Furthermore, the compliance rate of the treatment shall be calculated through the counting of the vials given back by the patient.

The patient shall be given new treatment, with the same code, enough until the next visit.

Visit 4 (Week 12)

In this visit the symptoms of the disease shall be valued with the two scales used in the study and the treatments that the patient has required during the 12 weeks following the end of the treatment under consideration.

Same as the first visit, they shall be asked to turn in a stool sample and they shall be taken a blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years old.
* Informed consent signed by the patient.
* Patients with Irritable Bowel Syndrome diagnosed by Roma IV criteria

Exclusion Criteria:

* Patients who took antibiotics until two weeks prior to study.
* Patients who have taken other probiotics two months prior.
* Patients with other intestinal inflammatory diseases.
* Pregnant, breastfeeding or patients who do not compromise to use an efficient contraceptive method during the development of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline on IBS-SSS (Irritable Bowel Syndrome-Severity Scoring System) scale at 4, 8 and 12 weeks | 12 weeks
  IBS index measures the severity of the disease, wich takes into account aspects such as pain, abdominal distension, intestinal habit and quality of life of the patient with IBS
  Categories of severity according to punctuation on the index IBS-SSS
  * Mild: 75 <175
  * Moderate: 175 <300
  * Severe: > 300

SECONDARY OUTCOMES:
Change from baseline on IBS-QoL (Irritable Bowel Syndrome-Quality of Life) index at 4, 8 and 12 weeks | 12 weeks
  IBS-QoL measures the impact of the disease on the quality of life of patients with IBS
  The questionnaire consists of 34 questions with a score of 1 to 5 in each of them.
Change from baseline on values of hemogram to final visit | 12 weeks
  Complete blood count
Change from baseline on values of blood glucose to final visit | 12 weeks
  Blood glucose parameters (mg/dL)
Change from baseline on values of blood sodium to final visit | 12 weeks
  Blood sodium parameters (mEq/L)
Change from baseline on values of blood potassium to final visit | 12 weeks
  Blood potassium parameters (mEq/L)
Change from baseline on values of blood chlorine to final visit | 12 weeks
  Blood chlorine parameters (mEq/L)
Change from baseline on values of blood creatinine to final visit | 12 weeks
  Blood creatinine parameters (mg/dL)
Change from baseline on values of blood HDL, LDL and total cholesterol to final visit | 12 weeks
  Blood HDL, LDL an total cholesterol parameters (mg/dL)
Change from baseline on values of blood triglycerides to final visit | 12 weeks
  Blood triglycerides parameters (mg/dL)
Change from baseline on values of blood C-reactive protein to final visit | 12 weeks
  Blood C-reactive protein parameters (mg/L)
Change from baseline on values of blood gamma glutamyl transferase (GGT) to final visit | 12 weeks
  Blood GGT parameters (mg/L)
Change from baseline on values of blood glutamic pyruvic transaminase (GPT) to final visit | 12 weeks
  Blood GPT parameters (mg/L)
Gut microbiota changes from baseline to final visit | 12 weeks
  Alpha Diversity, Beta Diversity, and Composition, Using R16s Gene Sequencing of a Stool Sample
Compliance rate at 4, 8 and 12 12 weeks | 12 weeks
  Assess compliance rate at each visit

OTHER OUTCOMES:
Adverse events on weeks 4, 8 and 12 | 12 week
  Number of adverse events reported by the patient at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Navarro López, PhD; MD, Principal Investigator — Universidad Católica San Antonio de Murcia (UCAM). MiBioPath Group.
Locations (1):
- MiBioPath UCAM, Murcia, Spain